CLINICAL TRIAL: NCT00771498
Title: An Evaluation of the Pharmacological Interaction of Lopinavir 800mg - Ritonavir 200mg Combination and Rifampin in Subjects Presenting Tuberculosis, With Contraindication for Antiretroviral Regimens Including Efavirenz
Brief Title: An Evaluation of the Pharmacological Interaction of Lopinavir/r and Rifampin
Acronym: A06-295
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Valeria Cavalcanti Rolla, Head of Laboratorio de Pesquisa Clinica em Micobacterioses, IPEC, Oswaldo Cruz Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: A06-295
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infection; Tuberculosis
Keywords: rifampin; lopinavir; drug interaction; pharmacokinetic
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lopinavir (Other): Patients with HIV/TB co-infection will receive treatment for both infection, and PK of lopinavir 800mg + ritonavir 200mg (PO BID) during 5 months will be performed
  Interventions: Drug: Lopinavir

INTERVENTIONS:
Drug: Lopinavir — ARV treatment: 2 NRTIs + lopinavir/r 800mg / 200 mg (4 tablets of Kaletra) every 12 hours, daily and orally Antituberculosis treatment: rifampin (600 mg/daily) + isoniazide (400 mg/daily) for 6 months, both in fasting condition + pirazinamide (2000 mg) for the first two months
  Other Names: Kaletra

SUMMARY:
This is a pharmacokinetic, descriptive, open-label, prospective, multicentric, national study in Aids and tuberculosis co-infected patients, to be laboratory and clinically monitored during the treatment with lopinavir-ritonavir and rifampin medications.

Study population: Thirty patients older than 18 years, both male and female, which present active tuberculosis and failure or contraindication for any motive to an efavirenz will be selected to participate in the study.

Objectives:

* Evaluate the pharmacokinetics of lopinavir-800mg / ritonavir-200mg combination (every 12 h) in association with rifampin-containing anti-tuberculosis regimens, in patients presenting tuberculosis and HIV-infected with indication to antiretroviral treatment according to Brazilian Ministry of Health's guidelines, with contraindication to the use of NNTRI.
* Describe the adverse events observed during the tuberculosis treatment period with rifampin associated with antiretroviral therapy consisting of lopinavir-800mg / ritonavir-200mg every 12 hours.
* Describe clinical, immunological and virological endpoints throughout the study with these drugs.

DETAILED DESCRIPTION:
Some attempts have been made to evaluate the pharmacokinetics of lopinavir using ritonavir as booster by some researchers with dosages of 400/100 and 533/133 mg (the last dosage would be achieved with an additional capsule of lopinavir/ritonavir) but the results were disappointing because AUC was importantly decreased with the introduction of rifampin in both situations (BERTZ et al, 2000).

La Porte et al (2004) presented the results of a pharmacokinetic study using two other dosage regimens, lopinavir-400mg/ritonavir-400mg and lopinavir-800mg/ritonavir-200mg co-administered with rifampin in healthy volunteers. With both doses, AUCs were reestablished, using an increased dose of only ritonavir, or a doubled dose of lopinavir/ritonavir. However, the minimum plasma concentration with the combination of lopinavir 800mg-ritonavir 200mg was lower in some timepoints than that recommended to achieve a good virologic effect. The reported adverse events, such as headache, nausea, diarrhea, fatigue and abdominal pain/cramps, were similar in both arms. However, there was a higher rate of liver toxicity in the lopinavir-400mg/ritonavir-400mg dose arm, with grade 2/3 ALT/SGTP elevations occurring in 5 subjects compared to 2 subjects in the lopinavir-800mg/ritonavir-200mg dose arm. Virological suppression was not evaluated because this was a pharmacokinetic study in healthy volunteers. In this case, liver toxicity might be explained by higher ritonavir doses, and strategies that can reduce the ritonavir dosage to permit a lower incidence of liver toxicity and other gastrointestinal events would be of extreme practical utility.

Recently, both WHO (WHO, 2003) and CDC (MMWR, 2004) recommend lopinavir 400mg-ritonavir 400mg every 12 hours in combination with rifampin in countries with limited resources, based solely in this study in healthy volunteers (La PORTE, 2004). In spite of the significant contribution to the knowledge on interaction among those drugs, this study does not reproduce the reality in clinical practice, because the volunteers were healthy, antiretroviral and anti-tuberculosis regimens were not given in full doses and lopinavir-ritonavir were introduced first and rifampin was added only after 14 days. In clinical practice, tuberculosis treatment is the priority (BRASIL, Ministério da Saúde, 2006), and the antiretroviral regimen is started later, after a period of at least 30 days, in order to observe tolerability and adverse events that usually occurs within the first month of tuberculosis treatment (PEDRAL-SAMPAIO 1997).

The scientific community reacted with surprise to this recommendation because there was no evidence in HIV-infected patients, that antiretroviral drugs and rifampin combination is as safe as described in healthy volunteers, as well as the concern about the frequency of adverse events that may occur with this combination. Furthermore, efforts have not been made to establish evidence that can support the use of a potent antiretroviral agent within the context of rescue regimens, among HAART-experienced patients. The perspective of another therapeutic possibility that may be used concomitantly with rifampin as a rescue medication in HIV-infected patients presenting tuberculosis and who have failed to antiretroviral regimen may represent the only option. Therapeutic regimens for tuberculosis without rifampin are less efficient, extend the negative baciloscopy, are associated with the biggest mortality besides being longer (1 year) and use an injectable drug during the first 3 months (streptomycin). Because lopinavir is a drug with an increased genetic barrier to resistance (MENDOZA & SORIANO, 2004) it may represent an excellent therapeutic option for patients who do not have other antiretroviral alternative.

In Brazil, the current marketed soft gel capsule formulation of Kaletra (lopinavir/ritonavir) presents some limitations such as the need for refrigeration and a moderately elevated incidence rate of diarrhea as an adverse event, between 25 to 28%, both among antiretroviral naïve and experienced patients (MURPHY et al, 2005; FEINBERG et al, 2000). Recently, the FDA (Food and Drug Administration, EUA) approved a new Kaletra (lopinavir/ritonavir) tablet formulation. The new formulation is based on a Meltrex™ (melt extrusion) technology, which requires no refrigeration (AWNI et al, 2005). Kaletra (lopinavir/ritonavir) tablets showed a lower incidence of diarrhea, in a pharmacokinetic study in healthy volunteers, when compared to other results found in studies that used the soft gel capsules (17.4%) (KLEIN et al, 2005). This scenario seems favourable for countries like Africa, where a refrigerator is a limitant condition for patients and treatment sites. A strategy of using tablets, without additional ritonavir seems promising.

Taking into account: (1) the complexity of the coinfection tuberculosis-HIV and the limited treatment options for both infections, as well as an urgent need to evaluate new options of antiretroviral regimens; (2) The results of La Porte et al (2004), that developed a pharmacokinetic study in which a pharmacokinetic drug interaction of two different doses of lopinavir/ritonavir co-administered with rifampin (600 mg/day) were evaluated; and (3) the pharmacokinetic study presented by Awni et al (2005), that showed pharmaceutic equivalence between Kaletra(lopinavir/ritonavir) soft gel capsules and tablets; we propose a clinical study in TB-HIV coinfected subjects using the association of lopinavir-ritonavir tablets and rifampin to evaluate its pharmacokinetics and safety.

This study may benefit patients co-infected with TB/HIV, particularly those with advanced immunodeficiency and who have shown failure to antiretroviral regimens including efavirenz or who may have any contraindication to their use (hypersensitivity or intolerance).

Thirty patients older than 18 years, both male and female, which present active tuberculosis and failure or contraindication for any motive to an efavirenz will be selected to participate in the study.

Antiretroviral treatment will consist of two NRTIs in combination or associated with a nucleotide analogue (tenofovir) and a combination of lopinavir-800 mg and ritonavir-200 mg (4 tablets of Kaletra) every 12 hours, daily and orally. A genotyping during screening will be conducted in order to optimize the combination therapy.

Antituberculosis treatment will consist on rifampin (600 mg/daily) isoniazide and (400 mg/daily), both in fasting condition and for 6 months; and pirazinamide (2.000 mg) for the first two months, according to the Ministry of Health recommendations. Doses will be adjusted for subjects who weight less than 45 kg. For patients who will be re-treated for tuberculosis, etambutol will be added in a dose of 1.200 mg/daily during the 6-month treatment. Those patients who need the use of any alternative regimen (without rifampin) will be excluded from study. In case of occurrence of gastrointestinal intolerance to rifampin, this one may be used after breakfast, but these data should be recorded in the patient chart in order to correlate it with pharmacokinetics data.

Lopinavir-Ritonavir should be started after 1 month after the beginning of antituberculosis treatment, at the visit of 30 days. The Lopinavir-Ritonavir dosage will be titrated during the first week of treatment, as follows:

1. on Days 30, 31 and 32: patients will receive lopinavir-ritonavir 400/100 mg (2 tablets) every 12 hours.
2. On Days 33, 34 and 35: patients will receive lopinavir-ritonavir 600/150 mg (3 tablets) every 12 hours.
3. From Day 36 until day 180: patients will receive lopinavir-ritonavir 800/200mg (4 tablets) every 12 hours, unless reduced on day 60 (refer to section 14.6).

After 6 months of tuberculosis treatment, if the patient fulfills the clinical and bacteriological criteria for cure, the antituberculosis drugs will be withdrawn and lopinavir-ritonavir (Kaletra®) will be maintained. However, the dose of Kaletra® (lopinavir/ritonavir) will be reduced to lopinavir 400mg / ritonavir 100mg (2 tablets) every 12 hours.

BERTZ A; HSU W; LAM L; ET AL. Pharmacokinetics interactions between Kaletra and other non HIV drugs. 5th International Congress on drug therapy in HIV infection. Glasgow UK October 22-26 2000. Poster 438.

BRASIL, MINISTÉRIO DA SAÚDE, 2006. Recomendações para o tratamento de adultos e adolescentes infectados pelo virus HIV.

EINBERG J, BRUN S, MARSS T, KING M, BENSON C, DEEKS S, KESSLER H, MURPHY R, GULICK R, WHEELER D, HICKS C, ERON J, SAX P, STRYKER R, RIDDLER S, THOMPSON M, REAL K, HSU A, BERTZ R, KEMPF D, JAPOUR A, SUN E. Durable Suppression of HIV+ RNA After Two Years of Kaletra (ABT-378/ritonavir) Therapy in Single Protease Inhibitor Experienced Patients. 5th International Congress on Drug Therapy in HIV Infection, Glasgow, UK (October 22-26, 2000)

LA PORTE CJL; COLBERS EPH; BERTS ET AL. Pharmacokinetics of adjusted-dose lopinavir-ritonavir combined with rifampin in healthy volunteers. Antimicrob. Agents Chemother 48:1553-1560 2004

MMWR Updated guidelines for the use of rifamycins for the treatment of tuberculosis among HIV-infected patients taking protease inhibitors or Nonnucleoside reverse transcriptase inhibitors, version 1.20.2004

MENDOZA, C. & SORIANO, V. Resistance to HIV protease inhibitors: mechanisms and clinical consequences. Curr. Drug Metab., 5(4):321-8, 2004.

MURPHY R, DA SILVA B, McMILLAN F, HICKS C, ERON J, WOLFE P, GULICK R, GLESBY M, THOMPSON M, BENSON C, WHITE AC, ALBRETCH M, KESSLER H, NIEMI K, KING K, CALHOUN D, KING M, HANNA G, BRUN S. Seven Year Follow-up of a Lopinavir/ritonavir (LPV/r)-Based Regimen in Antiretroviral (ARV)-Naïve Subjects. 10th EACS, Dublin 2005. Poster PE7.9/3.

PEDRAL-SAMPAIO DB, NETTO EM, ALCÂNTARA AP, SOUZA J, MOURA L, BRITES C ET AL. Use of Standard Therapy for Tuberculosis is Associated with Increased Adverse Reactions in Patients with HIV. BJID, 1(3): 123-130, 1997;

WHO (WORLD HEALTH ORGANIZATION). Scaling up antiretroviral therapy in resource-limited settings. Guidelines for a public health approach, 2003.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, with HIV infection and an active tuberculosis diagnosis. Women must have a negative pregnancy test and use a birth control method (barrier or Depo-Provera contraceptive) throughout the study and at investigator's discretion considered as reliable. To guarantee the security of the volunteers the pregnancy test in urine will be repeated to each visit.
* Patients who present contraindication for NNRTI use. Contraindication may be obtained through a history of virologic resistance (prior use of efavirenz with comproved virologic failure in a subject with good adherence), genotyping test indicative of mutations that provide resistance to these drugs, intolerance, or hypersensitivity.
* Patients must be older than 18 years.
* HIV infection documented by two positive ELISA tests for HIV and one confirmatory test (immunoblot or immunofluorescence), which may be replaced by a plasma VL using Roche-PCR test, Chiron Branched DNA or NASBA (BioMerrieux).
* The tuberculosis diagnostic can be proved through one positive culture with identification of M. tuberculosis. Besides, a patient will be eligible if he/she presents clinical signs and symptoms suggestive of tuberculosis, the radiological aspects are compatible, and other oportunistic deseases are excluded, even if specimen baciloscopy is negative, according to Brazilian Guidelines (BRASIL, Ministério da Saúde, 2004);
* Patients who do not require the use of medications with established contraindication for concomitant use with lopinavir-ritonavir, such as: amiodarone, astemizole, bepridil, bupropione, cisapride, clorazepate, clozapim, diazepam, encainide, flecainide, flurazepam, meperidine, midazolam, primozide, piroxicam, propafenone, propoxifeno, quinidine, rifabutin, terfenadine, triazolam, zolpidem, dihydroergotamine and ergotamine.
* Patient agrees not to use any medication (even herbal medications or natural products) without previous knowledgement and consent from investigator throughout the study. Patient also agrees to notify the investigator of any medication that has been changed (started or replaced) during the study.
* Patients should date and sign volunteer the informed consent before entering in the study and after a full explanation of the study nature. If the patient is unable, his/her legally authorized representative will sign on his/her behalf.

Exclusion Criteria:

* Patient has a previous history of hypersensitivity or known resistance or acquired to rifampin or to lopinavir-ritonavir.

  2. Evidence of toxic substances abuse, such as alcohol and/or illicit drugs (Attachment B).
* Viral B and/or C hepatitis co-infection.
* Patient presents one or more abnormalities in the following blood laboratory tests: STGO and/or STGP and/or alkaline phosphatase > 5,1 fold upper normal limit, or bilirrubin > 1.5 mg/dl. If the patient is not eligible at this moment due the risk of hepatotoxicity, an alternative treatment for tuberculosis will be offered (according to the recommendations of the Ministry of Health) in order to reduce the risk of serious hepatopaty and to allow the use of any concomitant antiretroviral scheme. This patient will be excluded of the study, but he will be able to be treated and accompanied in the responsible sites for the study up to the end of the tuberculosis treatment if it is the wish of the patient.
* Documented genotypic resistance to lopinavir/ritonavir on the screening sample.
* In the investigator's opinion, patient predicts a low compliance to the proposed study according to the clinical history for a given subject.
* Patient with history of prior use of Kaletra® (lopinavir, ritonavir) with comproved virologic or genotypic failure or serious intolerance needing change of antiretroviral treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Plasma levels of rifampin and lopinavir-ritonavir (pharmacokinetics). | 15, 45 and 180 days post-study treatment start

SECONDARY OUTCOMES:
HIV response to treatment | 90 and 180 days post-study treatment start
Adverse events | Each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Valeria C Rolla, PhD, Principal Investigator — Oswaldo Cruz Foundation; Valeria C Rolla, PhD, Study Chair — Oswaldo Cruz Foundation
Locations (3):
- Brazil (3):
  - University of Espirito Santo, Vitória, Espírito Santo
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC), Rio de Janeiro, Rio de Janeiro
  - Instituto Oswaldo Cruz (IOC), Rio de Janeiro, Rio de Janeiro